CLINICAL TRIAL: NCT01851369
Title: A Phase I/II Trial of TRC102 (Methoxyamine HCl) in Combination With Temozolomide in Patients With Relapsed Solid Tumors and Lymphomas
Brief Title: TRC102 and Temozolomide for Relapsed Solid Tumors and Lymphomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alice Chen, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130118; 13-C-0118
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Lymphomas; Solid Tumors; NSCLC; Metastatic Colon Carcinoma; Granulosa Cell Ovarian Cancer
Keywords: Solid Tumors; Lymphomas; DNA Damage; Pharmacodynamics; Pharmacokinetics
MeSH Terms: conditions — Lymphoma; Colonic Neoplasms | interventions — methoxyamine; Tomography, X-Ray Computed; atropine sulfate-diphenoxylate hydrochloride drug combination; Prochlorperazine; Metoclopramide; Serotonin 5-HT3 Receptor Antagonists; Serotonin; Aprepitant; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Treatment with Oral methoxyamine hydrochloride (TRC102) and oral Temozolomide (TMZ) (Experimental): Combination treatment with oral methoxyamine hydrochloride (TRC102) and oral Temozolomide (TMZ) for days 1-5 of 28-day cycles.
  Interventions: Drug: TRC102; Diagnostic Test: CT scan; Other: Lomotil; Other: Prochlorperazine; Other: Metoclopramide; Other: 5-HT3 antagonist; Other: Aprepitant; Procedure: Biopsy

INTERVENTIONS:
Drug: TRC102 — Methoxyamine hydrochloride (TRC102) has been shown to potentiate the activity of temozolomide by preventing base excision repair (BER) and allowing cleavage of TRC102 bound deoxyribonucleic acid (DNA), which will cause DNA strand breaks in cancer cells. We hypothesize that oral TRC102 can be safely co-administered with Temozolomide (TMZ) and would potentiate DNA damage caused by TMZ resulting in antitumor responses.
  Other Names: Methoxyamine hydrochloride
Diagnostic Test: CT scan — CT scans will be performed at baseline, and repeat scans will be performed every 2 cycles (every 3 cycles for participants on study more than one year).
  Other Names: Computed tomography
Other: Lomotil — If diarrhea develops and does not have an identifiable cause other than study drug administration, anti-diarrheal's such as Lomotil (diphenoxylate hydrochloride (HCl) 2.5 mg + atropine sulfate 0.025 mg/tablet) dosed according to package insert or loperamide 4 mg by mouth (po) after the first unformed stool with 2 mg po every 2 hours as long as unformed stools continue (4 mg every 4 hours while asleep). No more than 16 mg of loperamide should be taken in during a 24-hour period.
  Other Names: Diphenoxylate hydrocholoride
Other: Prochlorperazine — If a participant develops nausea/vomiting, an anti-emetic such as prochlorperazine may be given.
  Other Names: Compro
Other: Metoclopramide — If a participant develops nausea/vomiting, an anti-emetic such as metoclopramide may be given.
  Other Names: Reglan
Other: 5-HT3 antagonist — If a participant develops nausea/vomiting, an anti-emetic such as 5-HT3 antagonist may be given.
  Other Names: 5-hydroxytryptamine
Other: Aprepitant — If a participant develops nausea/vomiting, an anti-emetic such as aprepitant may be given.
  Other Names: Emend
Procedure: Biopsy — Tumor biopsies will be optional during the escalation phase.

SUMMARY:
Background:

- Methoxyamine hydrochloride (TRC102) is a new cancer treatment drug that may help improve the results of chemotherapy. It blocks tumor cells' attempts to repair damaged deoxyribonucleic acid (DNA), which may allow chemotherapy to kill the cells more easily. Researchers want to see how well it works with temozolomide, a chemotherapy drug that is designed to damage tumor cell DNA. These drugs will be given to people who have advanced solid tumors or lymphomas that have not responded to earlier treatments.

Objectives:

- To test the safety and effectiveness of TRC102 and temozolomide for advanced solid tumors and lymphomas.

Eligibility:

- Individuals at least 18 years of age who have advanced solid tumors or lymphomas that have not responded to earlier treatments.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Tumor samples may also be collected. The size and location of the tumors will be determined with imaging studies.
* Participants will take TRC102 and temozolomide for 28-day cycles of treatment. They will take temozolomide and TRC 102 by mouth once a day on days 1-5. Participants will keep a diary to record doses and any side effects.
* Treatment will be monitored with frequent blood tests and imaging studies. Tumor samples will also be collected.
* Participants will continue their treatment as long as the cancer does not grow and there are no severe side effects.

DETAILED DESCRIPTION:
Background:

* Base excision repair (BER) of deoxyribonucleic acid (DNA) repair pathway has been implicated in resistance to both alkylating and antimetabolite chemotherapy.
* TRC102 (methoxyamine hydrochloride (HCl) acts through a novel mechanism to inhibit BER and has demonstrated the ability to potentiate the activity of the alkylating agent temozolomide (TMZ), in vitro and in vivo. We hypothesize that TRC102 can be safely co-administered with TMZ and would potentiate DNA damage caused by TMZ, resulting in antitumor responses.
* Based on responses measured during the Phase I portion of the trial, we will further explore the efficacy of this combination in patients with metastatic colon carcinoma, non-small cell lung cancer (NSCLC), and granulosa cell ovarian cancer

Primary Objective:

* To establish the safety, tolerability, and maximum tolerated dose (MTD) of oral TRC102 in combination with oral TMZ in patients with refractory solid tumors
* Evaluate the pharmacokinetic (PK) profile of oral TRC102 when administered in combination with TMZ.
* To explore the response rate of this combination in patients with colon cancer, NSCLC, and granulosa cell ovarian cancer

Secondary Objective:

-To explore the progression free survival rate of this combination in patients with colon cancer, NSCLC, and granulosa cell ovarian cancer

Exploratory Objectives:

* Investigate tumor genomic and transcriptomic alterations potentially associated with sensitivity and/or the development of resistance to TRC102 and temozolomide.
* Determine the effects of the study treatment on the level of histone gamma-H2A histone family member X (H2AX) in circulating tumor cells (CTCs) and tumor and correlate the gamma-H2AX response in tumor and CTCs
* Determine the effects of the study treatment on the levels of cleaved caspase 3, epithelial- mesenchymal transition, and abdominoperineal excision (APE) in tumor and CTCs
* Determine and characterize the effects of study treatment on erythrocytes
* Characterize the clinical presentation of hemolysis observed in earlier study subjects and explore the possible mechanisms

Eligibility:

* Phase I: histologically confirmed solid tumors that have progressed on standard therapy known to prolong survival or for which no standard treatment options exist
* Phase II: histologically confirmed adenocarcinoma of the colon post at least two lines of therapy, NSCLC post at least two lines of therapy, or granulosa cell ovarian cancer post at least one line of therapy
* No major surgery, radiation, or chemotherapy within 4 weeks prior to entering the study
* Adequate organ function
* Healthy adult volunteers greater than or equal to 18 years of age will be consented to donate research blood

Please note: healthy adult volunteers will no longer be recruited to provide blood for this study as we will no longer perform the hemolysis analysis.

Study Design: Phase I

* This is an open-label Phase I trial; traditional 3+3 design.
* Oral TRC102 and oral TMZ will be administered daily, days 1-5 in 28-day cycles
* Once the MTD is established, up to 15 additional patients will be enrolled at the MTD to further evaluate that dose for PK and pharmacodynamic (PD) endpoints for evidence of DNA damage and apoptosis.
* During the escalation phase, tumor biopsies will be optional. During the expansion phase, (once MTD is reached), mandatory paired tumor biopsies will be pursued in the 15 additional patients enrolled to further evaluate progressive disease (PD) endpoints.

Phase II

* This is a 3-arm Simon 2-stage design trial evaluating independently the response rate of patients with colon, NSCLC, and granulosa cell ovarian cancer.
* Patients with a body surface area (BSA) of greater than or equal to 1.6 m(2) will receive 125 mg of TRC 102 and 150 mg/m(2) of TMZ PO qday x 5 every 28 days (DL6). Patients with a BSA of <1.6 m(2) will receive 100 mg of TRC 102 and 150 mg/m(2) of TMZ by mouth (PO) every (q)day x 5 every 28 days (Dose Level (DL)5). Each cycle will be 28 days.
* The accrual ceiling for the Phase II portion is 75 patients.
* Mandatory paired tumor biopsies will be pursued to further evaluate PD endpoints.

ELIGIBILITY:
* Eligibility Criteria (Patients)
* Phase I: histologically confirmed solid tumors that have progressed on standard therapy known to prolong survival or for which no standard treatment options exist.
* Phase II: histologically confirmed colorectal adenocarcinoma post at least two lines of therapy, non-small cell lung cancer (NSCLC) post at least two lines of therapy, or granulosa cell ovarian cancer post at least one line of therapy. Patients must have measurable disease.
* Age greater than18 years. Because no dosing or adverse event data are currently available on the use of methoxyamine hydrochloride (TRC102) in combination with Temozolomide (TMZ) in patients less than 18 years of age, children are excluded from this study.
* Patients enrolling in the expansion cohorts must have disease amenable to biopsy and be willing to undergo pre-and post-treatment biopsies.
* Eastern Cooperative Oncology Group (ECOG) performance status less than 2 (Phase I), less than or equal to 1(Phase II).
* Life expectancy of greater than 3 months
* Patients must have normal organ and marrow function as defined below:
* Absolute neutrophil count greater than 1,500/mcL
* Hemoglobin greater than or equal to 10 g/dL without transfusion within 1 week prior to enrollment

Platelets greater than or equal to 100,000/mcL

Total bilirubin less than or equal to1.5 X institutional ULN

Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/alanine transaminase (ALT) serum glutamic-pyruvic transaminase (SGPT)(SGPT) less than or equal to 3 X institutional upper limit of normal; 5.0 x upper limit of normal (ULN) in cases of liver metastases

creatinine less than or equal to 1.5 X institutional ULN

OR

creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels greater than 1.5 mg/dL

-The effects of study drug on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for at least 3 months after dosing with study drugs ceases. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of study drug administration.

* Patients must have completed any chemotherapy, radiation therapy, or biologic therapy greater than or equal to 4 weeks (or 5 half-lives, whichever is shorter) prior to entering the study (6 weeks for nitrosoureas or mitomycin C). Patients must be greater than or equal to 2 weeks since any prior administration of a study drug in a Phase 0 or equivalent study and greater than or equal to 1 week from palliative radiation therapy. Patients must have recovered to eligibility levels from prior toxicity or adverse events. Treatment with bisphosphonates is permitted.
* Patients must be able to swallow whole tablets or capsules; nasogastric or gastric (G)-tube administration is not allowed.
* Ability to understand and the willingness to sign a written informed consent document and to undergo tumor biopsies in the expansion phase.

Exclusion Criteria (Patients)

* Patients who are actively receiving any other investigational agents.
* Patients with active brain metastases or carcinomatous meningitis are excluded from this clinical trial. Patients with treated brain metastases, whose brain metastatic disease has remained stable for greater than or equal to 4 weeks without requiring steroid and anti-seizure medications are eligible to participate.
* Phase II only: No other prior malignancies are allowed except for the following:

  * Adequately managed stage 0 (carcinoma in situ), I, or II basal cell or squamous cell carcinoma from which the patient is currently in complete remission.
  * Any other cancer from which the patient has been disease-free for three years.
  * Adequately managed stage I or II well differentiated thyroid or prostate cancer is also eligible, wherein the patient is not required to be in complete remission.
* Phase II only: patients with colorectal cancer with known MSI-high disease who have not previously been treated with immunotherapy or who have refused treatment with immunotherapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TRC102 or TMZ.
* Uncontrolled intercurrent illness including, but not limited to, serious untreated infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because the effects of the study drugs on the developing fetus are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study drugs, breastfeeding should be discontinued prior to the first dose of study drug and women should refrain from nursing throughout the treatment period and for 3 months following the last dose of study drug.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of possible pharmacokinetic (PK) interactions with TRC102.

(Healthy volunteer blood donors)

Please note: healthy adult volunteers will no longer be recruited to provide blood for this study as we will no longer perform the hemolysis analysis.

* Age greater than 18 years; hemoglobin greater than or equal to 12 g/dL; no history of bleeding problems; not taking aspirin or any medication that may affect erythrocyte biochemistry
* Willingness to sign the healthy volunteer informed consent form.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-07-12 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Requests for all collected individual participant data (IPD) data from clinical trials, conducted under a binding collaborative agreement between National Cancer Institute (NCI/Division of Cancer Treatment and Diagnosis (DCTD) and a pharmaceutical/biotechnology company, that are not under data safety monitoring board (DSMB) monitoring must be in compliance with the terms of the binding collaborative agreement and must be approved by NCI/DCTD and the Pharmaceutical Collaborator (i.e., the NCI Experimental Therapeutics Clinical Trials Network (ETCTN) Director in conjunction with the NCI/DCTD Regulatory Affairs Branch).

REFERENCES:
- [Background] Liu L, Nakatsuru Y, Gerson SL. Base excision repair as a therapeutic target in colon cancer. Clin Cancer Res. 2002 Sep;8(9):2985-91. PMID 12231545
- [Background] Yan L, Bulgar A, Miao Y, Mahajan V, Donze JR, Gerson SL, Liu L. Combined treatment with temozolomide and methoxyamine: blocking apurininc/pyrimidinic site repair coupled with targeting topoisomerase IIalpha. Clin Cancer Res. 2007 Mar 1;13(5):1532-9. doi: 10.1158/1078-0432.CCR-06-1595. PMID 17332299
- [Background] Kinders RJ, Hollingshead M, Lawrence S, Ji J, Tabb B, Bonner WM, Pommier Y, Rubinstein L, Evrard YA, Parchment RE, Tomaszewski J, Doroshow JH; National Cancer Institute Phase 0 Clinical Trials Team. Development of a validated immunofluorescence assay for gammaH2AX as a pharmacodynamic marker of topoisomerase I inhibitor activity. Clin Cancer Res. 2010 Nov 15;16(22):5447-57. doi: 10.1158/1078-0432.CCR-09-3076. Epub 2010 Oct 5. PMID 20924131
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-C-0118.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase (Ph) 1 Dose Level -2 Methoxyamine (TRC102) 25mg & Temozolomide (TMZ) 75mg/m^2: No participants were enrolled in this group. Cycle = 28 days; Methoxyamine (TRC102) 25mg by mouth (PO) everyday (QD) on days 1-5; Temozolomide (TMZ) 75mg/m^2 PO QD on days 1-5.
- Phase 1 Dose Level -1 Methoxyamine (TRC102) 25mg & Temozolomide 100mg/m^2: No participants were enrolled in this group. Cycle = 28 days; Methoxyamine (TRC102) 25mg by mouth (PO) everyday (QD) on days 1-5; Temozolomide (TMZ) 100mg/m^2 PO QD on days 1-5.
- Phase 1 Solid Tumor Dose Level 1 Methoxyamine (TRC102) 125mg & Temozolomide 75mg/m^2: Cycle = 28 days; Methoxyamine (TRC102) 125mg by mouth (PO) everyday (QD) on days 1-5; Temozolomide (TMZ) 75mg/m^2 PO QD on days 1-5.
- Phase 1 Solid Tumor Dose Level 2 Methoxyamine (TRC102) 50mg & Temozolomide 125mg/m^2: Cycle = 28 days; Methoxyamine (TRC102) 50mg by mouth (PO) everyday (QD) on days 1-5; Temozolomide (TMZ) 125mg/m^2 PO QD on days 1-5.
- Phase 1 Solid Tumor Dose Level 3 Methoxyamine (TRC102) 50mg & Temozolomide 150mg/m^2: Cycle = 28 days; Methoxyamine (TRC102) 50mg by mouth (PO) everyday (QD) on days 1-5; Temozolomide (TMZ) 150mg/m^2 PO QD on days 1-5.
- Phase 1 Solid Tumor Dose Level 4 Methoxyamine (TRC102) 75mg & Temozolomide 150mg/m^2: Cycle = 28 days; Methoxyamine (TRC102) 75mg by mouth (PO) everyday (QD) on days 1-5; Temozolomide (TMZ) 150mg/m^2 PO QD on days 1-5.
- Phase 1 Solid Tumor Dose Level 5 Methoxyamine (TRC102) 100mg & Temozolomide 150mg/m^2: Cycle = 28 days; Methoxyamine (TRC102) 100mg by mouth (PO) everyday (QD) on days 1-5; Temozolomide (TMZ) 150mg/m^2 PO QD on days 1-5.
- Phase 1 Solid Tumor Dose Level 6 Methoxyamine (TRC102) 125mg & Temozolomide 150mg/m^2: Cycle = 28 days; Methoxyamine (TRC102) 125mg by mouth (PO) everyday (QD) on days 1-5; Temozolomide (TMZ) 150mg/m^2 PO QD on days 1-5.
- Phase 1 Solid Tumor Dose Level 7 Methoxyamine (TRC102) 150mg & Temozolomide 150mg/m^2: Cycle = 28 days; Methoxyamine (TRC102) 150mg by mouth (PO) everyday (QD) on days 1-5; Temozolomide (TMZ) 150mg/m^2 PO QD on days 1-5.
- Phase 1 Solid Tumor Dose Level 8 Methoxyamine (TRC102) 150mg & Temozolomide 200mg/m^2: Cycle = 28 days; Methoxyamine (TRC102) 150mg by mouth (PO) everyday (QD) on days 1-5; Temozolomide (TMZ) 200mg/m^2 PO QD on days 1-5.
- Ph 2 Colorectal Cancer TMZ 150mg/m^2/Methoxyamine 125mgOR100mg(Based on Body Surface Area); Ph2 Non Small Cell Lung Cancer TMZ 150mg/m^2/Methoxyamine125mgOR100mg(Based on Body Surface Area); Ph 2 Granulosa Cell Temozolomide 150mg/m^2 & Methoxyamine 125mgOR 100mg (Based on Body Surface Area): Cycle = 28 days; Methoxyamine (TRC102) 125mg by mouth (PO) everyday (QD) on days 1-5; Temozolomide (TMZ) 150mg/m^2 PO QD on days 1-5 for participants with a body surface area (BSA) ≥ 1.6 m^2 OR Cycle = 28 days; Methoxyamine (TRC102) 100mg by mouth (PO) everyday (QD) on days 1-5; Temozolomide (TMZ) 150mg/m^2 PO QD on days 1-5 for participants with a body surface area (BSA) < 1.6 m^2.
Period: Phase I Dose Escalation
Arm/Group | Phase (Ph) 1 Dose Level -2 Methoxyamine (TRC102) 25mg & Temozolomide (TMZ) 75mg/m^2 | Phase 1 Dose Level -1 Methoxyamine (TRC102) 25mg & Temozolomide 100mg/m^2 | Phase 1 Solid Tumor Dose Level 1 Methoxyamine (TRC102) 125mg & Temozolomide 75mg/m^2 | Phase 1 Solid Tumor Dose Level 2 Methoxyamine (TRC102) 50mg & Temozolomide 125mg/m^2 | Phase 1 Solid Tumor Dose Level 3 Methoxyamine (TRC102) 50mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 4 Methoxyamine (TRC102) 75mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 5 Methoxyamine (TRC102) 100mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 6 Methoxyamine (TRC102) 125mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 7 Methoxyamine (TRC102) 150mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 8 Methoxyamine (TRC102) 150mg & Temozolomide 200mg/m^2 | Ph 2 Colorectal Cancer TMZ 150mg/m^2/Methoxyamine 125mgOR100mg(Based on Body Surface Area) | Ph2 Non Small Cell Lung Cancer TMZ 150mg/m^2/Methoxyamine125mgOR100mg(Based on Body Surface Area) | Ph 2 Granulosa Cell Temozolomide 150mg/m^2 & Methoxyamine 125mgOR 100mg (Based on Body Surface Area)
Started | 0 | 0 | 3 | 6 | 4 | 8 | 3 | 3 | 5 | 3 | 0 | 0 | 0
Completed | 0 | 0 | 3 | 6 | 4 | 7 | 3 | 3 | 5 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Declined to participate (before treatment started) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase I Maximum Tolerated Dose Expansion
Arm/Group | Phase (Ph) 1 Dose Level -2 Methoxyamine (TRC102) 25mg & Temozolomide (TMZ) 75mg/m^2 | Phase 1 Dose Level -1 Methoxyamine (TRC102) 25mg & Temozolomide 100mg/m^2 | Phase 1 Solid Tumor Dose Level 1 Methoxyamine (TRC102) 125mg & Temozolomide 75mg/m^2 | Phase 1 Solid Tumor Dose Level 2 Methoxyamine (TRC102) 50mg & Temozolomide 125mg/m^2 | Phase 1 Solid Tumor Dose Level 3 Methoxyamine (TRC102) 50mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 4 Methoxyamine (TRC102) 75mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 5 Methoxyamine (TRC102) 100mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 6 Methoxyamine (TRC102) 125mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 7 Methoxyamine (TRC102) 150mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 8 Methoxyamine (TRC102) 150mg & Temozolomide 200mg/m^2 | Ph 2 Colorectal Cancer TMZ 150mg/m^2/Methoxyamine 125mgOR100mg(Based on Body Surface Area) | Ph2 Non Small Cell Lung Cancer TMZ 150mg/m^2/Methoxyamine125mgOR100mg(Based on Body Surface Area) | Ph 2 Granulosa Cell Temozolomide 150mg/m^2 & Methoxyamine 125mgOR 100mg (Based on Body Surface Area)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 10 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 10 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase II
Arm/Group | Phase (Ph) 1 Dose Level -2 Methoxyamine (TRC102) 25mg & Temozolomide (TMZ) 75mg/m^2 | Phase 1 Dose Level -1 Methoxyamine (TRC102) 25mg & Temozolomide 100mg/m^2 | Phase 1 Solid Tumor Dose Level 1 Methoxyamine (TRC102) 125mg & Temozolomide 75mg/m^2 | Phase 1 Solid Tumor Dose Level 2 Methoxyamine (TRC102) 50mg & Temozolomide 125mg/m^2 | Phase 1 Solid Tumor Dose Level 3 Methoxyamine (TRC102) 50mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 4 Methoxyamine (TRC102) 75mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 5 Methoxyamine (TRC102) 100mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 6 Methoxyamine (TRC102) 125mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 7 Methoxyamine (TRC102) 150mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 8 Methoxyamine (TRC102) 150mg & Temozolomide 200mg/m^2 | Ph 2 Colorectal Cancer TMZ 150mg/m^2/Methoxyamine 125mgOR100mg(Based on Body Surface Area) | Ph2 Non Small Cell Lung Cancer TMZ 150mg/m^2/Methoxyamine125mgOR100mg(Based on Body Surface Area) | Ph 2 Granulosa Cell Temozolomide 150mg/m^2 & Methoxyamine 125mgOR 100mg (Based on Body Surface Area)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 16 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 16 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data was collected and is reported here for all 93/93 participants, including one participant on phase 1 dose level 4 who declined to participate (before treatment started).
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Solid Tumor Dose Level 1 Methoxyamine (TRC102) 125mg & Temozolomide 75mg/m^2 | Phase 1 Solid Tumor Dose Level 2 Methoxyamine (TRC102) 50mg & Temozolomide 125mg/m^2 | Phase 1 Solid Tumor Dose Level 3 Methoxyamine (TRC102) 50mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 4 Methoxyamine (TRC102) 75mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 5 Methoxyamine (TRC102) 100mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 6 Methoxyamine (TRC102) 125mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 7 Methoxyamine (TRC102) 150mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 8 Methoxyamine (TRC102) 150mg & Temozolomide 200mg/m^2 | Ph 2 Colorectal Cancer TMZ 150mg/m^2/Methoxyamine 125mgOR100mg(Based on Body Surface Area) | Ph2 Non Small Cell Lung Cancer TMZ 150mg/m^2/Methoxyamine125mgOR100mg(Based on Body Surface Area) | Ph 2 Granulosa Cell Temozolomide 150mg/m^2 & Methoxyamine 125mgOR 100mg (Based on Body Surface Area) | Total
Number analyzed (Participants) | 3 | 6 | 4 | 8 | 3 | 10 | 15 | 3 | 16 | 16 | 9 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 2 | 7 | 3 | 7 | 10 | 3 | 8 | 8 | 8 | 63
  >=65 years | 1 | 1 | 2 | 1 | 0 | 3 | 5 | 0 | 8 | 8 | 1 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.13 (12.22) | 57.82 (6.83) | 62.9 (14.03) | 58.54 (5.37) | 48.57 (11.52) | 58.44 (10.45) | 61.51 (11.25) | 57 (5.91) | 62.24 (10.75) | 61.97 (14.1) | 49.14 (18.4) | 59.11 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 4 | 2 | 5 | 6 | 2 | 5 | 4 | 9 | 43
  Male | 1 | 4 | 2 | 4 | 1 | 5 | 9 | 1 | 11 | 12 | 0 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 1 | 1 | 0 | 8
  Not Hispanic or Latino | 3 | 5 | 4 | 8 | 3 | 7 | 13 | 3 | 15 | 14 | 9 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 1 | 2 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 2 | 1 | 12
  White | 2 | 2 | 3 | 7 | 3 | 6 | 10 | 3 | 14 | 10 | 8 | 68
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 4 | 8 | 3 | 10 | 15 | 3 | 16 | 16 | 9 | 93

OUTCOME MEASURES:

1. Primary Outcome: Phase 2: Response Rate of This Combination in Participants With Colon Cancer, Non-small Cell Lung Cancer (NSCLC), and Granulosa Cell Ovarian Cancer
Description: Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on-study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions.
Time Frame: Response rate at one year
Population: A total of 41/93 participants were analyzed: 0/52 phase 1 participants were analyzed as this outcome measure was for the phase 2 participants only; 41/41 phase 2 participants were evaluable for response rate.
Measure: Count of Participants; unit: Participants
Arm/Group | Ph 2 Colorectal Cancer TMZ 150mg/m^2/Methoxyamine 125mgOR100mg(Based on Body Surface Area) | Ph2 Non Small Cell Lung Cancer TMZ 150mg/m^2/Methoxyamine125mgOR100mg(Based on Body Surface Area) | Ph 2 Granulosa Cell Temozolomide 150mg/m^2 & Methoxyamine 125mgOR 100mg (Based on Body Surface Area)
Number analyzed (Participants) | 16 | 16 | 9
Participants
  Complete Response | 0 | 0 | 0
  Partial Response | 1 | 0 | 0
  Stable Disease | 3 | 10 | 5
  Progressive Disease | 8 | 3 | 2
  Not Assessed Due to Death on Study | 1 | 0 | 0
  Not Assessed Due to Clinical Progression | 2 | 2 | 1
  Not Assessed Due to Refusing Further Treatment | 1 | 1 | 1

2. Primary Outcome: The Number of Dose Limiting Toxicities Observed in Participants Receiving Oral TRC102 in Combination With Oral TMZ
Description: Dose-limiting toxicities (DLTs) are defined as toxicities occurring within the first cycle of treatment felt to be possibly, probably, or definitely related to administration of study drugs and fulfilling one of the following criteria: Grade 4 neutropenia, febrile neutropenia, neutropenic infection: Grade ≥ 3 neutropenia with grade ≥ 3 infection, Grade ≥ 3 thrombocytopenia, a drop in hemoglobin (Hgb) ≥3.0 g/dL over one week, and all Grade ≥ 3 non-hematologic toxicity other than: non-bloody diarrhea Grade 3 that is corrected to Grade ≤ 2 within 24 hours, nausea and vomiting Grade 3 that is corrected to Grade ≤ 1 within 24 hours, creatinine Grade 3 corrected to Grade ≤ 1 within 48 hours, and Grade 3 electrolyte abnormalities. Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. And Grade 5 is death related to adverse event.
Time Frame: At dose-limiting toxicity (DLT) determined in the first cycle; approximately 28 days
Population: 36/37 participants in the phase I dose escalation cohort were analyzed because one participant in dose level 3 declined to participate (before treatment started).
Measure: Number; unit: Dose limiting toxicities
Arm/Group | Phase 1 Solid Tumor Dose Level 1 Methoxyamine (TRC102) 125mg & Temozolomide 75mg/m^2 | Phase 1 Solid Tumor Dose Level 2 Methoxyamine (TRC102) 50mg & Temozolomide 125mg/m^2 | Phase 1 Solid Tumor Dose Level 3 Methoxyamine (TRC102) 50mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 4 Methoxyamine (TRC102) 75mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 5 Methoxyamine (TRC102) 100mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 6 Methoxyamine (TRC102) 125mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 7 Methoxyamine (TRC102) 150mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 8 Methoxyamine (TRC102) 150mg & Temozolomide 200mg/m^2
Number analyzed (Participants) | 3 | 6 | 4 | 7 | 3 | 3 | 7 | 3
Dose limiting toxicities
  A Drop in Hemoglobin (Hgb) ≥3.0 g/dL Over One Week | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Grade 4 Neutropenia | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Grade 4 Thrombocytopenia | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

3. Primary Outcome: Phase 1 Pharmacokinetic (PK) Profile of Oral TRC102 When Administered in Combination With Temozolomide (TMZ) as Measured by Maximum Plasma Concentration (Cmax) of TRC102: Mean (Standard Deviation)
Description: Blood samples will be collected, and pharmacokinetics will be assessed in the phase I portion of the study. Samples will be analyzed using a validated LC-MS or LC-MS/MS method in human plasma. The maximum observed analyte concentration in plasma was reported.
Time Frame: First 5 days of treatment
Population: 51/52 participants were analyzed for plasma PK in phase 1 because one participant declined to participate (before treatment started).
Measure: Mean (Standard Deviation); unit: Micromolar (µM)
Arm/Group | Phase 1 Solid Tumor Dose Level 1 Methoxyamine (TRC102) 125mg & Temozolomide 75mg/m^2 | Phase 1 Solid Tumor Dose Level 2 Methoxyamine (TRC102) 50mg & Temozolomide 125mg/m^2 | Phase 1 Solid Tumor Dose Level 3 Methoxyamine (TRC102) 50mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 4 Methoxyamine (TRC102) 75mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 5 Methoxyamine (TRC102) 100mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 6 Methoxyamine (TRC102) 125mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 7 Methoxyamine (TRC102) 150mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 8 Methoxyamine (TRC102) 150mg & Temozolomide 200mg/m^2
Number analyzed (Participants) | 3 | 6 | 4 | 7 | 3 | 10 | 15 | 3
Micromolar (µM) | 0.75 (0.49) | 1.49 (1.07) | 0.97 (0.27) | 2.36 (2.68) | 3.51 (2.52) | 7.11 (8.21) | 7.45 (5.39) | 7.54 (5.40)

4. Primary Outcome: Phase 1 Pharmacokinetic (PK) Profile: the Percentage of TRC102 Dose Recovered From Participant Urine in Participants Treated With Oral TRC102 in Combination With Temozolomide (TMZ)
Description: Urine samples will be collected, and pharmacokinetics will be assessed in phase I portion of the study. Samples will be analyzed using a validated liquid chromatography-mass spectrometry (LC-MS) or liquid chromatography with tandem mass spectrometry (LC-MS-MS) method.
Time Frame: First day of treatment
Population: 51/52 participants were analyzed for urine PK in phase 1 because one participant declined to participate (before treatment started).
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Phase 1 Solid Tumor Dose Level 1 Methoxyamine (TRC102) 125mg & Temozolomide 75mg/m^2 | Phase 1 Solid Tumor Dose Level 2 Methoxyamine (TRC102) 50mg & Temozolomide 125mg/m^2 | Phase 1 Solid Tumor Dose Level 3 Methoxyamine (TRC102) 50mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 4 Methoxyamine (TRC102) 75mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 5 Methoxyamine (TRC102) 100mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 6 Methoxyamine (TRC102) 125mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 7 Methoxyamine (TRC102) 150mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 8 Methoxyamine (TRC102) 150mg & Temozolomide 200mg/m^2
Number analyzed (Participants) | 3 | 6 | 4 | 7 | 3 | 10 | 15 | 3
Percentage | 1.6 (1.2) | 0.8 (0.3) | 0.8 (0.5) | 2.5 (2.9) | 4.0 (3.1) | 4.8 (5.2) | 4.1 (4.6) | 3.8 (2.3)

5. Primary Outcome: Phase 1 Maximum Tolerated Dose (MTD) of Oral TRC102 in Participants With Refractory Solid Tumors.
Description: The MTD or recommended Phase II dose is the dose level at which no more than 1 of 6 participants experience dose-limiting toxicity (DLT) during the first cycle of treatment, and the dose below that at which at least 2 (of ≤ 6) participants have DLT as a result of the drug. DLTs are defined as toxicities occurring within the first cycle of treatment felt to be possibly, probably, or definitely related to administration of study drugs and fulfilling one of the following criteria: Grade 4 neutropenia, febrile neutropenia, neutropenic infection: Grade ≥ 3 neutropenia with grade ≥ 3 infection, Grade ≥ 3 thrombocytopenia, a drop in hemoglobin (Hgb) ≥3.0 g/dL over one week, and all Grade ≥ 3 non-hematologic toxicities other than: non-bloody diarrhea Grade 3 that is corrected to Grade ≤ 2 within 24 hours, nausea and vomiting Grade 3 that is corrected to Grade ≤ 1 within 24 hours, creatinine Grade 3 corrected to Grade ≤ 1 within 48 hours, and Grade 3 electrolyte abnormalities.
Time Frame: First cycle of treatment; approximately 28 days
Population: 51/52 participants were analyzed in phase 1 because one participant declined to participate (before treatment started).
Measure: Number; unit: mg
Groups:
- All Participants: All participants on phase I who received at least one dose of TRC102 and Temozolomide.
Arm/Group | All Participants
Number analyzed (Participants) | 51
mg | 125

6. Primary Outcome: Phase 1 Maximum Tolerated Dose (MTD) of Oral Temozolomide (TMZ) in Participants With Refractory Solid Tumors.
Description: The MTD or recommended Phase II dose is the dose level at which no more than 1 of 6 participants experience dose-limiting toxicity (DLT) during the first cycle of treatment, and the dose below that at which at least 2 (of ≤ 6) participants have DLT as a result of the drug. DLTs will be defined as toxicities occurring within the first cycle of treatment and is felt to be possibly, probably, or definitely related to administration of study drugs and fulfills one of the following criteria: hematologic toxicities - Grade 4 neutropenia, febrile neutropenia, neutropenic infection: Grade ≥ 3 neutropenia with grade ≥ 3 infection, Grade ≥ 3 thrombocytopenia, a drop in hemoglobin (Hgb) ≥3.0 g/dL over one week, any degree of lymphopenia, or leukopenia in the absence of grade 4 neutropenia will not be considered dose limiting, and Grade ≥ 3 non-hematologic toxicity. Grade ≥ 3 electrolyte abnormalities will not be considered dose limiting.
Time Frame: First cycle of treatment; approximately 28 days
Population: 51/52 participants were analyzed in phase 1 because one participant declined to participate (before treatment started).
Measure: Number; unit: mg/m^2
Arm/Group | All Participants
Number analyzed (Participants) | 51
mg/m^2 | 150

7. Secondary Outcome: Phase 2: Progression Free Survival Rate of This Combination in Participants With Colon Cancer, Non-small Cell Lung Cancer (NSCLC), and Granulosa Cell Ovarian Cancer
Description: Progression free survival rate of this combination in participants with colon cancer, NSCLC, and granulosa cell ovarian cancer. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) and is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum onstudy (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions.
Time Frame: Duration on study, an average of 130 days
Population: 41/41 participants in phase 2 were analyzed. 0/52 participants in phase 1 were analyzed as this was a Phase 2-specific outcome measure, thus the table reports data for phase 2 reporting groups only.
Measure: Median (Full Range); unit: Months
Arm/Group | Ph 2 Colorectal Cancer TMZ 150mg/m^2/Methoxyamine 125mgOR100mg(Based on Body Surface Area) | Ph2 Non Small Cell Lung Cancer TMZ 150mg/m^2/Methoxyamine125mgOR100mg(Based on Body Surface Area) | Ph 2 Granulosa Cell Temozolomide 150mg/m^2 & Methoxyamine 125mgOR 100mg (Based on Body Surface Area)
Number analyzed (Participants) | 16 | 16 | 9
Months | 1.97 [0.6 to 6.2] | 3.02 [1.2 to 15.1] | 5.52 [0.9 to 25.1]

8. Other Pre Specified Outcome: Phase 1 and Phase 2: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, an average of 115 days.
Population: 92/93 participants were analyzed because one participant in phase 1 dose level 3 declined to participate (before treatment started).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Solid Tumor Dose Level 1 Methoxyamine (TRC102) 125mg & Temozolomide 75mg/m^2 | Phase 1 Solid Tumor Dose Level 2 Methoxyamine (TRC102) 50mg & Temozolomide 125mg/m^2 | Phase 1 Solid Tumor Dose Level 3 Methoxyamine (TRC102) 50mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 4 Methoxyamine (TRC102) 75mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 5 Methoxyamine (TRC102) 100mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 6 Methoxyamine (TRC102) 125mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 7 Methoxyamine (TRC102) 150mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 8 Methoxyamine (TRC102) 150mg & Temozolomide 200mg/m^2 | Ph 2 Colorectal Cancer TMZ 150mg/m^2/Methoxyamine 125mgOR100mg(Based on Body Surface Area) | Ph2 Non Small Cell Lung Cancer TMZ 150mg/m^2/Methoxyamine125mgOR100mg(Based on Body Surface Area) | Ph 2 Granulosa Cell Temozolomide 150mg/m^2 & Methoxyamine 125mgOR 100mg (Based on Body Surface Area)
Number analyzed (Participants) | 3 | 6 | 4 | 7 | 3 | 10 | 15 | 3 | 16 | 16 | 9
Participants | 3.0 | 6 | 4 | 7 | 3 | 10 | 15 | 3 | 16 | 16 | 9

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, an average of 115 days.
Description: 92/93 participants were analyzed because one participant in phase 1 dose level 3 declined to participate (before treatment started).
Arm/Group | Phase 1 Solid Tumor Dose Level 1 Methoxyamine (TRC102) 125mg & Temozolomide 75mg/m^2 | Phase 1 Solid Tumor Dose Level 2 Methoxyamine (TRC102) 50mg & Temozolomide 125mg/m^2 | Phase 1 Solid Tumor Dose Level 3 Methoxyamine (TRC102) 50mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 4 Methoxyamine (TRC102) 75mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 5 Methoxyamine (TRC102) 100mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 6 Methoxyamine (TRC102) 125mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 7 Methoxyamine (TRC102) 150mg & Temozolomide 150mg/m^2 | Phase 1 Solid Tumor Dose Level 8 Methoxyamine (TRC102) 150mg & Temozolomide 200mg/m^2 | Ph 2 Colorectal Cancer TMZ 150mg/m^2/Methoxyamine 125mgOR100mg(Based on Body Surface Area) | Ph2 Non Small Cell Lung Cancer TMZ 150mg/m^2/Methoxyamine125mgOR100mg(Based on Body Surface Area) | Ph 2 Granulosa Cell Temozolomide 150mg/m^2 & Methoxyamine 125mgOR 100mg (Based on Body Surface Area)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/4 | 0/7 | 0/3 | 2/10 | 2/15 | 0/3 | 1/16 | 0/16 | 1/9
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/6 | 2/4 | 1/7 | 1/3 | 4/10 | 9/15 | 2/3 | 9/16 | 9/16 | 2/9
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 4/4 | 7/7 | 3/3 | 10/10 | 15/15 | 3/3 | 16/16 | 16/16 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Solid Tumor Dose Level 1 Methoxyamine (TRC102) 125mg & Temozolomide 75mg/m^2 (N=3) | Phase 1 Solid Tumor Dose Level 2 Methoxyamine (TRC102) 50mg & Temozolomide 125mg/m^2 (N=6) | Phase 1 Solid Tumor Dose Level 3 Methoxyamine (TRC102) 50mg & Temozolomide 150mg/m^2 (N=4) | Phase 1 Solid Tumor Dose Level 4 Methoxyamine (TRC102) 75mg & Temozolomide 150mg/m^2 (N=7) | Phase 1 Solid Tumor Dose Level 5 Methoxyamine (TRC102) 100mg & Temozolomide 150mg/m^2 (N=3) | Phase 1 Solid Tumor Dose Level 6 Methoxyamine (TRC102) 125mg & Temozolomide 150mg/m^2 (N=10) | Phase 1 Solid Tumor Dose Level 7 Methoxyamine (TRC102) 150mg & Temozolomide 150mg/m^2 (N=15) | Phase 1 Solid Tumor Dose Level 8 Methoxyamine (TRC102) 150mg & Temozolomide 200mg/m^2 (N=3) | Ph 2 Colorectal Cancer TMZ 150mg/m^2/Methoxyamine 125mgOR100mg(Based on Body Surface Area) (N=16) | Ph2 Non Small Cell Lung Cancer TMZ 150mg/m^2/Methoxyamine125mgOR100mg(Based on Body Surface Area) (N=16) | Ph 2 Granulosa Cell Temozolomide 150mg/m^2 & Methoxyamine 125mgOR 100mg (Based on Body Surface Area) (N=9)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (6) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Infections and infestations - Other, covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — progressive disease death
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Pneuomonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Solid Tumor Dose Level 1 Methoxyamine (TRC102) 125mg & Temozolomide 75mg/m^2 (N=3) | Phase 1 Solid Tumor Dose Level 2 Methoxyamine (TRC102) 50mg & Temozolomide 125mg/m^2 (N=6) | Phase 1 Solid Tumor Dose Level 3 Methoxyamine (TRC102) 50mg & Temozolomide 150mg/m^2 (N=4) | Phase 1 Solid Tumor Dose Level 4 Methoxyamine (TRC102) 75mg & Temozolomide 150mg/m^2 (N=7) | Phase 1 Solid Tumor Dose Level 5 Methoxyamine (TRC102) 100mg & Temozolomide 150mg/m^2 (N=3) | Phase 1 Solid Tumor Dose Level 6 Methoxyamine (TRC102) 125mg & Temozolomide 150mg/m^2 (N=10) | Phase 1 Solid Tumor Dose Level 7 Methoxyamine (TRC102) 150mg & Temozolomide 150mg/m^2 (N=15) | Phase 1 Solid Tumor Dose Level 8 Methoxyamine (TRC102) 150mg & Temozolomide 200mg/m^2 (N=3) | Ph 2 Colorectal Cancer TMZ 150mg/m^2/Methoxyamine 125mgOR100mg(Based on Body Surface Area) (N=16) | Ph2 Non Small Cell Lung Cancer TMZ 150mg/m^2/Methoxyamine125mgOR100mg(Based on Body Surface Area) (N=16) | Ph 2 Granulosa Cell Temozolomide 150mg/m^2 & Methoxyamine 125mgOR 100mg (Based on Body Surface Area) (N=9)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (4)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 5 (8) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 2 (3) | 1 (1) | 1 (2) | 0 (0) | 3 (8) | 6 (8) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (2) | 2 (3) | 1 (1) | 4 (4) | 1 (1) | 2 (4) | 7 (10) | 0 (0) | 3 (3) | 4 (6) | 3 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 3 (7) | 4 (10) | 4 (7) | 2 (2) | 8 (18) | 10 (20) | 3 (19) | 12 (16) | 8 (16) | 6 (12)
Anorexia (Metabolism and nutrition disorders) | 2 (6) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 6 (6) | 5 (5) | 0 (0) | 3 (3) | 6 (7) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 3 (4) | 1 (2) | 2 (2) | 1 (1) | 5 (9) | 5 (10) | 1 (2) | 4 (5) | 1 (1) | 1 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 4 (6) | 1 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 3 (4) | 10 (14) | 2 (2) | 5 (6) | 5 (6) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 3 (4)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 2 (3) | 2 (2) | 3 (3) | 4 (9) | 1 (1) | 5 (6) | 5 (9) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (4) | 0 (0) | 2 (2) | 5 (5) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (2) | 2 (7) | 3 (5) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 3 (7) | 3 (4) | 3 (8)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 2 (4)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 4 (5) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 4 (4) | 4 (4) | 5 (11)
Dizziness (Nervous system disorders) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 5 (5) | 0 (0) | 3 (6) | 1 (1) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 1 (1) | 2 (3) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, right scleral irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (4) | 0 (0) | 3 (6) | 3 (3) | 1 (1) | 4 (5) | 2 (2) | 0 (0) | 6 (6) | 9 (16) | 4 (7)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 3 (6) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flashing lights (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Gastrointestinal disorders - Other, hypersalivation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, night sweat (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haptoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (3) | 2 (4) | 1 (2) | 3 (3) | 0 (0) | 2 (2) | 3 (7) | 1 (1) | 2 (2) | 4 (6) | 2 (3)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 3 (4)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hoarseness (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (15) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 3 (3) | 2 (4) | 1 (12)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (3) | 6 (15) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 4 (8) | 0 (0) | 8 (14) | 4 (7) | 4 (8)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (5) | 1 (1) | 2 (2) | 5 (7) | 10 (15) | 2 (2) | 10 (14) | 7 (9) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 2 (3) | 3 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (2) | 3 (4) | 0 (0) | 2 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 4 (6) | 3 (5)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 2 (5) | 0 (0) | 2 (2) | 3 (7) | 5 (6) | 2 (3) | 5 (10) | 7 (14) | 4 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 3 (3) | 1 (1) | 5 (6) | 2 (3) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Investigations - Other, LDH increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 2 (3) | 3 (6) | 3 (8) | 2 (2) | 6 (14) | 10 (19) | 3 (15) | 10 (19) | 11 (24) | 2 (11)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (4) | 6 (8) | 3 (9) | 6 (7) | 2 (3) | 5 (6) | 10 (27) | 3 (7) | 7 (9) | 11 (22) | 8 (14)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (8) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 3 (4) | 1 (1) | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (3) | 2 (2) | 2 (3) | 4 (6) | 0 (0) | 2 (2) | 6 (9) | 3 (10) | 5 (17) | 3 (6) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (3) | 4 (4) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Chest congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 3 (6) | 0 (0) | 2 (3) | 3 (7) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (6) | 4 (5) | 3 (3) | 4 (4) | 2 (3) | 3 (5) | 7 (11) | 1 (3) | 3 (3) | 7 (15) | 5 (5)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Weight loss (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 2 (3) | 4 (8) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 2 (12) | 1 (2) | 0 (0) | 1 (1) | 4 (11) | 3 (7) | 0 (0) | 2 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT01851369/Prot_SAP_000.pdf
  • Informed Consent Form: Cohort Treatment Consent (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT01851369/ICF_001.pdf
  • Informed Consent Form: Healthy Blood Donor Consent (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/69/NCT01851369/ICF_002.pdf
  • Informed Consent Form: Standard Phase I Consent (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT01851369/ICF_003.pdf